CLINICAL TRIAL: NCT07240948
Title: Functional Improvement in Subacute/Chronic Stroke Patients Through a Non-invasive Virtual-reality Based Telerehabilitation Home System
Brief Title: Functional Improvement in Subacute/Chronic Stroke Through Non-invasive Virtual-reality-Based Telerehabilitation
Acronym: MUVITY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Nora Therapeutics, Inc. (Industry); Muvity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS(AG)034/2025(6497); PI23/01680 (Other Grant/Funding Number: Fundación Instituto de Investigación Salud Carlos III)
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; chronic stroke rehabilitation; tele-rehabilitation; telestroke; telehealth; home rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open trial with blind evaluation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUVITY arm (Experimental): Users of the Muvity telerehabilitation system. At baseline, a therapist will elaborate a personalized treatment plan consisting of exercises and games to be carried out during 12 weeks in the patient's home. Muvity will be provided to each participant for the duration of the program (software of non-immersive virtual reality (niVR) through a depth camera installed in a personal computer (PC)). The user will see the exercises and serious games in the loaned PC as daily quests, in a gamified environment, to be completed in 30 min, three times per week. Alerts will be sent through Nora to remind the scheduled treatment, and a contact from the case-manager will be performed if the patient does not perform treatment. Questions about pain feeling perception and emotional wellbeing will be asked before and after each session automatically by the system and the patient will be able to contact the case manager/physiotherapist for questions/comments, and to receive feedback.
  Interventions: Device: Non- immersive virtual reality (niVR)-based telerehabilitation home program
- Control arm (No Intervention): Conventional at-home rehabilitation treatment and routine follow-up. The participant will receive an informative sheet with the description of the exercises prescribed by the physiatrist and elaborated by the physiotherapist, with the instructions to perform sessions of 30 min three times a week. The exercises will cover similar movements as the ones formulated in the telerehabilitation system for the intervention group. In the Nora app, the patient in the control group will need to actively report the timing of his/her rehabilitation treatment, and the same questions about pain feeling perception and emotional wellbeing before and after each treatment. However, no feedback of rehabilitation progress will be provided.

INTERVENTIONS:
Device: Non- immersive virtual reality (niVR)-based telerehabilitation home program — Muvity (software of non-immersive virtual reality (niVR) through a depth camera installed in a personal computer (PC)) will be provided with a personalized treatment plan to be carried out 3times/week along 12w in the patient's home. The user will see exercises and serious games as daily quests, in a gamified environment with alerts to remind the scheduled treatment. The potential exercises include following a virtual avatar to perform individual movements (shoulder flexion-extension, shoulder vertical or horizontal abduction-adduction, elbow flexion-extension, hip flexion-extension or hip abduction-adduction), squats or medio-lateral movements of the pelvis to control the body weight transfer. The serious games are oriented toward performing movements in activities of daily living, such as cooking, cleaning a mirror, or acting as a goalkeeper, or collecting apples.
  Arms: MUVITY arm

SUMMARY:
Stroke is the leading cause of disability in adults worldwide. Rehabilitation after a stroke is crucial, even after the acute phase: initially, it aims to recover the deficits caused by the stroke, but in the subacute/chronic phases the objective is to maintain the functional abilities already acquired. After the acute phase, traditional rehabilitation methods usually include exercises prescribed by a therapist that the patient performs on their own. However, their effectiveness is limited due to the lack of supervision, adherence, and insufficient information provided to the patient about their progress, which would require regular in-person contact with the patient. To date, public health systems have been unable to provide this kind of access to rehabilitation for post-stroke patients, with the risk of worsening deficits and a decline in quality of life. We plan to develop an individualized home-based monitoring program enhanced by telerehabilitation based on non-immersive virtual reality (without the need for VR goggles or other "gadgets") (MUVITY) for patients who suffered a stroke in the subacute/chronic phase.

Patients seen during an outpatient consultation who require rehabilitation will be randomly assigned either the usual treatment (they will receive a document describing the exercises to perform and a suggested schedule, togheter with an app for communication and health-education, Nora) or the MUVITY treatment: patients will be provided with the telerehabilitation system using a computer and camera where they will perform the rehabilitation exercises, which will be individually adapted according to their progress by a physiotherapist, together with Nora. We believe that MUVITY will lead to improved motor function, emotional well-being, and quality of life, increasing adherence to rehabilitation treatment compared with usual care, and that it can be used in terms of patient satisfaction and pain levels.

Our findings could confirm that telerehabilitation improves motor function and quality of life after stroke. Furthermore, since it is a home-based system, its use would considerably increase the number of patients who can receive treatment compared with in-person therapies, eliminating geographic barriers related to distance from rehabilitation centers and offering cost-effective access to effective treatment for all patients. Additionally, our system allows continuous interaction between patients and healthcare professionals, and provides information about their progress, which helps reduce stress related to uncertainty about the future and supports key aspects of monitoring patients in the subacute/chronic phase of stroke such as risk factor control and early detection of complications.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years-old
* Ischemic or hemorrhagic stroke within 3 to 12 months before inclusion
* Inclusion modified Rankin scale 1 to 3
* Motor rehabilitation requirements defined by the stroke neurologist/physiatrist in the out-patient clinic
* Bipedal standing: capable of keeping on two feet for two minutes without using hand supports.

Exclusion Criteria:

* Technological abilities: patient and caregiver do not manage smartphone and computer
* Severe aphasia/ language barrier with patient/caregiver that impairs communication
* Severe cognitive impairment (dementia) that affects short- and medium-term memory.
* End-of-life- or life-threatening pathology with an estimated survival <1 year.
* Receiving intense physical therapy (rehabilitation with at least one face-to-face physical treatment/week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Median change in the Motor Fugl-Meyer and Berg Balance Scales | From baseline to the end of treatment period (12 weeks)
  Description: Comparison of the median change between treatment arms in the Fugl-Meyer and Berg Balance Scales evaluated before and after treatment. The measurement will be performed in the first visit to establish a baseline in both Muvity and control arms. At the end of the treatment, a face-to-face visit by a researcher (trained occupational therapist) blinded to the treatment group will be performed, and a new evaluation of the scales will be performed. The outcome will be evaluated by the Mann-Whitney U test and Rank Transformation ANCOVA.

SECONDARY OUTCOMES:
Adherence levels to prescribed rehabilitation protocols | At the end of the treatment period (12 weeks from baseline)
  Comparison of the adherence to the prescribed rehabilitation protocols in both the Muvity and control arms. For the evaluation, automatic system data will be collected in the Muvity software for the intervention group (descriptive, no comparison). To compare the adherence between arms, a specific questionnaire has been developed and will be administered to all patients. In addition, patients in the control group will be able to register their rehabilitation sessions in a new functionality created in the Nora app.
Improvement in the self-perceived health status and quality of life | Baseline (before treatment initiation) and end-visit (after 12 weeks)
  Comparison of the self-perceived health status and quality of life, together with pain perception during the rehabilitation treatment, in both the Muvity and control arms. In both arms, evaluation will be performed by the HRQoL(Health-Related Quality of Life), PROMIS-10 (Patient-Reported Outcomes Measurement Information System 10-Item), HADs (Hospital Anxiety and Depression Scale) and Pain-VAS (Visual Analog Scale) patient-reported outcome measurements. A baseline evaluation will be performed before treatment initiation, and a second one at the end of the treatment period. A comparison of the median scores in the different groups at the end of the study, adjusted by baseline, and a comparison of the change in the scores of each individual patient will be performed. The outcome will be evaluated by the Mann-Whitney U test and Rank Transformation ANCOVA.
User performance evaluation | After weeks 2 and 12 (end of study) from treatment initiation
  Tracking of user performance progression through in-game metrics (e.g., level scores, duration at week 2 and 12 of treatment) in the Muvity treatment arm.

OTHER OUTCOMES:
Patient's satisfaction and usability evaluation | End of the treatment period (after 12 weeks)
  Test of patients' satisfaction and usability of the Muvity program will be performed through a Picker test-like PREM (patient-reported experience measurement) administered to patients in the interventional group

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All anonymized clinical, functional dynamic and kinematic individual patient data (IPD) together with identifying metadata (with exception of those related with Muvity intellectual property)
Time Frame: The IPD will be available at the end of the clinical study (from February 2027) until February 2037
Access Criteria: Data will be shared through e-mail contact with the PI, upon reasonable request

REFERENCES:
- See also: Muvity web-page — https://muvity.cat/about.html
- See also: Nora web-page — https://www.nora.bio/